CLINICAL TRIAL: NCT03788005
Title: Impact of an Early Out-of-bed Paradigm in Postoperative Outcomes of Chronic Subdural Hematomas: GET-UP Randomized Prospective Trial
Brief Title: GET-UP Trial: Impact of an Early Out-of-bed Paradigm in Postoperative Outcomes of Chronic Subdural Hematomas
Acronym: GET-UP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Sérgio Sousa, Principal Investigator, Centro Hospitalar do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-176 (151-DEFI/150-CES)
Record Dates: First submitted 2018-12-19; First posted 2018-12-27 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic Subdural Hematoma; Bed rest; Early mobilization
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Early Ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Early mobilization as soon as possible, within a maximum of 12 hours post-surgery.
  Subdural drains will be closed when the patient is allowed to mobilize and will be open during a nocturnal period of 8 hours. Subdural drains will be removed past 48 hours of surgery.
  Interventions: Procedure: Early mobilization
- Control Group (No Intervention): Bed rest with head of bed at 0 degrees for 48h. Subdural drains will be removed past 48 hours of surgery.

INTERVENTIONS:
Procedure: Early mobilization — Early mobilization as soon as possible and within a maximum of 12 hours following burr hole craniostomy for chronic subdural hematomas.
  Arms: Intervention group

SUMMARY:
Compare rates of medical complications, recurrence and outcome in 2 randomized groups of patients with surgical chronic subdural hematomas. The intervention group will be assigned to early mobilization (within 12 hours of the surgical procedure). The control group will be assigned to bed rest for 48 hours.

DETAILED DESCRIPTION:
At Centro Hospitalar do Porto it is routinely used burr hole craniostomy with subdural drains and 48 hours of bed rest for the surgical treatment of chronic subdural hematomas. After 48 hours the subdural drains are removed and the patient is allowed to mobilize for the first time.

The aim of the present study is to conduct a prospective, randomized, controlled trial with an early mobilization protocol vs 48 hours bed rest to determine the best strategy to reduce postoperative complications and improve functional outcomes.

There will be 2 groups:

* Control group: bed rest 48 hours post-surgery with removal of subdural drains after this period.
* Intervention group: Early mobilization protocol: as early mobilization as possible, within a maximum of 12 hours following surgery, with progressive autonomization in the ward as tolerated by the patient. Mobilization time will be recorded. At the time of assuming an upright position the drains will be closed and will only be open again when the patient is in supine position (8 hours per day of supine position). Subdural drains will be removed after 48 hours, similar to the practice in the control group.

Primary End-Point:

• Number of medical complications. Medical complication is defined as any occurrence which merits additional tests or, preferentially, requires any form of medical treatment. This includes respiratory infections, urinary infections, wound infections, meningitis, deep vein thrombosis, pulmonary embolism, cerebral infarction or hemorrhage, syncope, among others.

Secondary End-Points:

* Recurrence rates. A recurrence is defined as any chronic subdural hematoma ipsilateral to that of the original hematoma if a surgical strategy needs to be pursued.
* Functional status (using both GOS-E and mRS). Timeframes considered will be pre-operative functional status, functional status at discharge, functional status at 3 months post-operative.
* Mortality rates.
* Recurrence free survival.
* Time to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Surgically drained chronic subdural hematomas (Burr hole craniostomy)
* > or equal to 18 years old

Exclusion Criteria:

* Previous neurosurgery
* Surgery for another pathology performed at the same time
* > 6h sedation post-surgery
* Any previous condition that makes early mobilization impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2022-08-05 (Estimated)

PRIMARY OUTCOMES:
Medical Complications | From date of randomization until 3 months post-randomization
  Infections, venous thromboembolism, seizures

SECONDARY OUTCOMES:
Recurrence | At 3 months follow-up
  Recurrence of a chronic subdural hematoma if surgical intervention is required
Post-operative Modified Rankin scale | At 3 months follow-up
  Modified Rankin Scale from 0 (free of symptoms) to a maximum of 6 (dead)
Survival | At 3 months follow-up
  Survival
Length of hospital stay | From date of randomization until clinical discharge up to 36 months
  Time to clinical discharge
Post-operative GOS-E scale | At 3 months follow-up
  GOS-E scale from 1 (dead) to a maximum of 8 (upper good recovery - resumption of normal life within the capacity work even if pre-injury status has not been achieved; any existing deficits are not disabling)

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Sousa, MD, Principal Investigator — Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar Universitário do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kurabe S, Ozawa T, Watanabe T, Aiba T. Efficacy and safety of postoperative early mobilization for chronic subdural hematoma in elderly patients. Acta Neurochir (Wien). 2010 Jul;152(7):1171-4. doi: 10.1007/s00701-010-0627-4. Epub 2010 Mar 25. PMID 20336332
- [Background] Brennan PM, Kolias AG, Joannides AJ, Shapey J, Marcus HJ, Gregson BA, Grover PJ, Hutchinson PJ, Coulter IC; British Neurosurgical Trainee Research Collaborative. The management and outcome for patients with chronic subdural hematoma: a prospective, multicenter, observational cohort study in the United Kingdom. J Neurosurg. 2017 Oct;127(4):732-739. doi: 10.3171/2016.8.JNS16134. Epub 2016 Nov 11. PMID 27834599
- [Derived] Pinto V, Sousa SA, Vaz da Silva F, Ribeiro da Costa T, Fernandes AP, Batata R, Noronha C, Monteiro Silva J, Ferreira S, Sobral S, Alves C, Rangel R, Calheiros A; GET-UP Trial Collaborators. GET-UP Trial 1-year results: long-term impact of an early mobilization protocol on functional performance after surgery for chronic subdural hematoma. J Neurosurg. 2023 Nov 10;140(5):1434-1441. doi: 10.3171/2023.8.JNS231509. Print 2024 May 1. PMID 37948693
- [Derived] Sousa S, Pinto V, Vaz da Silva F, Ribeiro da Costa T, Fernandes A, Batata R, Noronha C, Monteiro Silva J, Ferreira S, Sobral S, Alves C, Rangel R, Calheiros A; GET-UP Trial Collaborators. Impact of an early mobilization protocol on the reduction of medical complications after surgery for chronic subdural hematoma: the GET-UP Trial. J Neurosurg. 2023 Mar 17;139(3):854-863. doi: 10.3171/2023.2.JNS222262. Print 2023 Sep 1. PMID 36933251